CLINICAL TRIAL: NCT03349294
Title: Clinical Study of Biokinetic Model of Iodine-131 in Total(Near) Thyroidectomy Patients.
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 106132-F
Record Dates: First submitted 2017-10-20; First posted 2017-11-21 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2017-11

CONDITIONS: Thyroidectomy
Keywords: Thyroid; Thyroidectomy; Iodine; Biokinetic; Ablation
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thyroid cancer patients who have undergone total thyroidectomy, postoperative iodine 131 treatment to ablation residual thyroid tissue, is the current clinical practice. The effective half-life of the iodine 131 in the human body and in vivo exposure dose can be assessed by the in vivo kinetic model published by ICRP, but this model is based on standard healthy people and can not be corrected for patients undergoing total thyroidectomy.

In this study, the investigators will use the actual clinical data to revise the biokinetic model of iodine-131 in patients with total thyroidectomy.

DETAILED DESCRIPTION:
Methods Patients:All patients undergoing thyroidectomy and are about to be treated with iodine 131 30mCi will be invited to join the study. Exclusion with gastrointestinal surgery.

Preparation:The patient of this study, their medication and diet and other matters needing attention, are in accordance with the original to accept iodine -131 30mCi treatment of the standard treatment.

Imaging Protocol:After oral administration of iodine 131, patients must undergo whole body scan, for 1 hour, 4 hours, 24 hours, 48 hours, 72 hours, 168 hours, respectively. Image collection will use GE Infinia Hawkeye 4 SPECT / CT with high energy general purpose collimator. The imaging parameters use the original I-131 whole body scan protocol.

Expected results:Image data is further analyzed by MATLAB software to obtain iodine 131 in the body of individual organs of the biological half-life and path strength percentage. This analysis can revise the iodine -131 biokinetic model of patients with total thyroidectomy, providing more accurate calculations and subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing thyroidectomy and are about to be treated with iodine 131 30mCi will be invited to join the study.

Exclusion Criteria:

* Exclusion with gastrointestinal surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing thyroidectomy and are about to be treated with iodine 131 30mCi will be invited to join the study. Exclusion with gastrointestinal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The I-131 distributed among the internal organs after the dose administration can be thoroughly analyzed according to a revised MATLAB program. | After oral administration of iodine 131, patients must undergo whole body scan, for 1 hour, 4 hours, 24 hours, 48 hours, 72 hours, 168 hours, respectively.
  Image data is further analyzed by MATLAB software

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chun Huang, Principal Investigator
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan